

Approval Period 06/21/2022 - 06/20/2023

## CONSENT INFORMATION SHEET

Localized mHealth approach to boosting COVID-19 testing and vaccine literacy, access, and uptake among women with criminal legal system involvement

## Dr. Megha Ramaswamy

We are asking you to take part in a NIH RADx-UP\* research study about attitudes about Covid-19 through the University of Kansas Medical Center (KUMC). Participation is optional, and you may change your mind at any time.

The program will last for one year. We will deliver health information about Covid -19 through a textweb platform that you can access on your phone, on a home computer, at a public library, or wherever you usually use the internet. We will ask you to complete a survey before the text web program, 1 month after the completed program and 12 months after completion. We will also check in you every three months so that we can update your contact information. Only the Tri-City Covid Attitudes team, Duke University and the NIH will have access to this information. All of which will be stored on a secure computer.

We hope that the information we gain is useful in creating a different way of informing others about Covid-19. The survey questions may be personal, (i.e. – your knowledge and attitudes). You do not have answer any question with which you are not comfortable. When we write up or discuss the results of the study, we will not use any names or any other information that can identify you. What you say will have no impact on any services that you receive at the University of Kansas Medical Center.

Duke University will store data that does not identify you. If you choose to provide your zip code, then that data may be linked to other data using your zip code. Duke University will transfer these data to a secure NIH database. These data will not be able to identify you. Other researchers may use this data for future studies. We will not ask your permission before sharing this data as it will not identify you.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health (NIH). This protects the researchers from being forced to give out personal information about you for legal proceedings. This does not stop you from voluntarily releasing information about yourself or your participation in this research.

One exception to the Certificate is if you agree that we can give out research information that identifies you. Your information will be shared for the purposes listed in this consent form. Other exceptions are information we must report if we learn about child abuse or neglect or if we think you might harm yourself or others.

You will receive compensation for participation. You will get \$25 for completing the baseline survey and the text web program. A month after completion for the program, you will get \$50 for completion of a follow-up survey. 12 months after completion of the program, you will get \$50 for completing another follow-up survey. Every three months while you are in the study, we will also stay in touch with you to update your contact information. You will get paid \$10 each



for your 3-month, 6-month and 9-month check-ins. The total amount you could get if you participate in all parts of the study over one year is \$155. If you leave the study early, you will be paid only for the visits you completed.

For our Kansas City and Birmingham participants, you will be on the same ClinCard that you have previously established. If you are in Oakland, you will continue to receive cash payments.

The KUMC Research Institute will be given your name, address, social security number, and the title of this study to allow them to set you up in the ClinCard system. Study payments are taxable income. A Form 1099 will be sent to you and the Internal Revenue Service if your payments are \$600 or more in a calendar year. a valid social security number or tax identification number, 30% of your payments will be set aside by KUMC and sent to the IRS for withholding on your behalf. Your participation in our study will not exceed \$600.

Your personal information will be kept on a secure computer. It will be removed from the computer after the study is over and the money on the card has been used. Your information will not be shared with other businesses. It will be kept completely confidential.

If you have questions about this study, please contact Dr. Megha Ramaswamy at 913-588-1053. For questions about your rights as a research participant, you may contact the KUMC Institutional Review Board (IRB) at (913) 588-1240 or <a href="mailto:IRBhelp@kumc.edu">IRBhelp@kumc.edu</a>.

If you want to be a part of this study, we ask that you provide your verbal consent. You will be mailed a

copy of this form to keep for your records. You will have the option of sharing or not sharing any identifiable information with the study.

Sincerely,

Sherri Anderson <u>sanderson10@kumc.edu</u> 913-205-1818

## \*WHAT ARE THE NIH AND RADX-UP?

The NIH stands for the National Institutes of Health. The NIH supports health research, including the RADx-UP program.

RADx-UP stands for Rapid Acceleration of Diagnostics - Underserved Populations. RADx-UP is a COVID19 research program.

